CLINICAL TRIAL: NCT03794739
Title: Ruolo Del Marcatore TMEM219 in Corso di Diabete di Tipo 1
Brief Title: Role of TMEM219 Marker in Type 1 Diabetes
Acronym: NPOD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Paolo Fiorina, MD, Professor of Endocrinogy University of Milan, Director of Endocrinology and Diabetology Unit ASST Fatebenefratelli-Sacco, University of Milan
Other Study IDs: 2018/ST/080
Record Dates: First submitted 2018-12-31; First posted 2019-01-07 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes mellitus; Beta cell loss; Beta cell apoptosis
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Serum, pancreatic sections, pancreatic islets.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Healthy subjects: Healthy subjects without diabetes, no recent surgery interventions, no malignancies no pregnancy.
  No intervention. No age limit.
- T1D individuals: Type 1 diabetic individuals with at least 3-year of duration of the disease. No recent surgery interventions, no malignancies no pregnancy.
  No intervention. No age limit.
- T2D individuals: Type 2 diabetic individuals with at least 5-year duration of the disease. No recent surgery interventions, no malignancies no pregnancy.
  No intervention. No age limit.
- AutoAb+ individuals: Individuals at risk for type 1 diabetes, with one or more autoantibody detected. No recent surgery interventions, no malignancies no pregnancy.
  No intervention. No age limit.

SUMMARY:
Type 1 diabetes (T1D) is a chronic metabolic disease characterized by autoimmune destruction of β cells of the insulin producing pancreatic islets. The different immunological approaches implemented to date to treat T1D have obtained a negligible number of insulin-independent individuals. The initial stages of diabetic disease are characterized by the massive and progressive infiltration of T cells and autoantibodies within the tissue with the consequent development of insulitis and subsequently, the destruction of pancreatic beta cells. The onset of T1D has been mainly associated to a dysregulation of the immune response. However, data are emerging on the importance of non-immunological factors responsible for the damage to pancreatic beta cells. The investigators have recently shown that the expression of the TMEM219 death factor is an essential factor in controlling the fate of stem cells in diabetes.

The aim of the study is to identify new markers in the mechanism of damage to pancreatic beta cells in the onset of type 1 diabetes, with particular reference to apoptotic factors such as TMEM219.

DETAILED DESCRIPTION:
METHODS OF RECRUITING THE SUBJECTS Healthy subjects, individuals with type 1 and type 2 diabetes and those who are at risk of developing diabetes will be enrolled. Enrollment was approved by the University of Florida Ethics Committee within the NPOD project, Network for the Pancreatic Organ Donors with Diabetes.

Duration of the study: 5 years.

EXPERIMENTAL PROCEDURE:

The following analyses will be performed on the collected and received samples:

* Study of TMEM219 expression and of other TMEM219-related markers by immunohistochemistry and immunofluorescence and western blot
* Study of TMEM219 expression and of other TMEM219-related markers by molecular biology analysis
* Analysis of the proteomic profile on collected biological liquids The above analyses will be performed at the Pediatric Clinical Research Center Romeo ed Enrica Invernizzi at the Sacco Hospital - University of Milan.

PREVIOUS EXPERIENCES The investigatore expertise in manipulating / studying the signaling involved in the pathogenesis of type 1 diabetes has been widely recognized in several publications in recent years (Diabetes 2013, Diabetes 2014, Diabetes 2015, Science Translational Medicine 2017) as well as the characterization of marker expression including TMEM219 (Cell Stem Cell 2015).

RELEVANCE OF THE STUDY The study offers the possibility to acquire new information on the pathogenesis of diabetes and to identify new target mechanisms for designing innovative therapeutic strategies in the treatment of diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Reported in the NPOD protocol

Exclusion Criteria:

* Reported in the NPOD protocol

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study already approved at the local Ethical Committee provides for the enrollment of the following groups of subjects:
  * subjects affected by diabetes (type 1, type 2, MODY)
  * subjects at risk of developing diabetes (positive screening for autoantibodies)
  * subjects not affected by diabetes Enrollment is coordinated by the University of Florida as part of the NPOD project, Network for the Pancreatic Organ Donors with Diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-08-08 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Altered TMEM219 expression in pancreatic islets/beta cells in diabetes. | 1-24 months
  Change of TMEM219 expression in pancreatic islets/beta cells of healthy subjects as compared to that of individuals with type 1 diabetes (T1D), with type 2 diabetes (T2D) and of those at risk for developing the disease.

SECONDARY OUTCOMES:
Increased beta cell loss due to a dysregulated TMEM219 signaling in diabetes. | 25 months-48 months
  Change in TMEM219-related factors and signaling in pancreatic islets/beta cells of healthy subjects as compared to individuals with T1D, with T2D and of individuals at risk for developing the disease.
Altered TMEM219-peripheral regulating factors in diabetes. | 49 months-60 months
  Change of peripheral factors involved in controlling TMEM219 expression/activation detected in the serum of healthy subjects as compared to individuals with T1D, with T2D and at risk for developing the disease.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Fiorina, MD, PhD, Principal Investigator — University of Milan
Locations (1):
- Pediatric Clinical Research Center, Milan, Italy